CLINICAL TRIAL: NCT03520309
Title: CARies DEtection in Children 03 - The Impact of Two Different Clinical Criteria for the Evaluation of Caries Lesions Around Restorations in Primary Teeth
Brief Title: Clinical Criteria for the Evaluation of Caries Lesions Around Restorations in Primary Teeth (CARDEC-03)
Acronym: CARDEC-03
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Fausto Medeiros Mendes, Associate professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: CARDEC-03
Record Dates: First submitted 2018-03-06; First posted 2018-05-09 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Dental Caries; Secondary Dental Caries
Keywords: Diagnosis; Visual inspection; Quality of Life; Restorations
MeSH Terms: conditions — Dental Caries; Disease | interventions — Dental Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- International Dental Federation (Experimental): Dental Treatment: according to the decision based on the International Dental Federation (FDI) criteria
  Interventions: Procedure: Dental treatment
- Caries Around Restorations System (Experimental): Dental Treatment: according to the decision based on the Caries Around Restorations System (CARS) and treatment decision proposed by the International Caries Classification and Management System (ICCMS)
  Interventions: Procedure: Dental treatment

INTERVENTIONS:
Procedure: Dental treatment — Treatment of all dental restorations of the children according to the diagnosis criteria

SUMMARY:
There is still great divergence in the aspects related to caries lesions around restorations. The methods and the systems used for the detection of secondary caries lesions have presented low validity. Also, the consequent treatment decisions of this kind of lesions have presented a lot of variation. However, the correct diagnosis of secondary caries may guarantee greater longevity to the restorative treatment, as well as oral health to the patients, reducing the cost and clinical time of the dentists. Therefore, the investigators aimed to perform this study to evaluate and compare two visual criteria for the evaluation of restorations in primary teeth in medium and long term outcomes for the patients, through a randomized clinical study. These criteria are the system proposed by the World Dental Federation (FDI) and the International Caries Classification and Management System - ICCMS.

DETAILED DESCRIPTION:
Among the available diagnosis criteria to detect caries lesions around restorations, there are the World Dental Federation (FDI) criteria and the International Caries Classification and Management System - ICCMS. However, few studies have evaluated the accuracy of both methods. The impact of the use of these methods in the treatment decisions regarding the restorations was also not evaluated. In relation to the detection of caries lesions around restorations in primary teeth, no randomized clinical study was performed, so the aim of this study is to establish the best diagnosis and treatment decision to caries around restorations in children. For this, three different studies will be carried out according the following specific aims: (1) to evaluate the accuracy of the FDI criteria and the system proposed by the ICCMS for the evaluation of caries lesions around restorations in primary teeth through a cross-sectional study design; (2) to evaluate the impact and cost of using these two criteria in treatment decisions related to the evaluation of restorations in primary teeth through a cross-sectional study design; (3) to evaluate the influence of the use of these two criteria for the evaluation of restorations in primary teeth in medium and long term outcomes for the patients, through a randomized clinical trial. To reach these objectives 626 restorations will be evaluated in children from 3 to 10 years who have looked for dental treatment in our dental school. They will be randomly allocated in two groups according to the diagnostic strategy used for caries detection around restorations: diagnosis and treatment decision based on the criteria of the International Dental Federation (FDI) (control group) or diagnosis and treatment decision based on the CARS detection criteria and treatment decision proposed by the ICCMS (experimental group). The consequent treatment decision of the restorations will be divided into no restorative intervention; repair or replacement of the restorations. Children will be treated by dentists, blinded to the criteria used to reach the treatment decision and then, will be monitored for two years. Reassessments will be performed by a blind examiner in relation to the child's allocation group, and the occurrence of outcomes will be assessed according to predefined criteria described for evaluation of restorations performed in the context of atraumatic restorative treatment. The primary outcome will be the need for restorative intervention during the follow-up of the restorations evaluated by the different criteria. This outcome is composed of several components. The reference standard will be the presence of caries lesion adjacent to the restoration after removal of the restoration, and their occurrence will be compared among the methods by survival analysis.

ELIGIBILITY:
Inclusion Criteria:

* Children who sought dental treatment in our dental school (School of Dentistry, University of Sao Paulo, Sao Paulo, Brazil)
* Children aged 3 to 6 years
* Children with at least one restoration on a primary tooth of any material, on any dental surface and regardless of its condition.

Exclusion Criteria:

* Children whose parents refuse to participate of the research
* Children who refuse to participate of the research or exhibited behavioral problems during the initial appointment
* All child's restorations will be included in the evaluation, except for restorations presenting fistula, abscess, pulp exposure, history of spontaneous dental pain or mobility.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 163 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Restoration survival | 24 months
  Major failures of restorations: restorations presenting failures that need replacement or teeth with pulp involvement, pain or that need extraction (except due to orthodontic reasons). For restorations involving occlusal surfaces, score 4 of Frencken et al. criteria (1996) will be considered. For restorations involving other surfaces, the scores 21, 30, and 40.
  The primary outcome was changed due to the COVID-19 pandemic situation. As we were not able to assess patients' restorations at 24 months, we could not evaluate the need for operative treatment at this time. Therefore, restoration survival was set as the primary outcome, as we can determine the restoration failure by the assessment date.

SECONDARY OUTCOMES:
Operative treatment needs of the evaluated restorations (success of restoration) | 24 months.
  The necessity to repair the evaluated restorations during the follow-up examinations will be assessed by the Roeleveld et al. (1996) criteria (scores 11, 12, 13 and 30) or Frencken et al. (1996) criteria (scores 2 and 3). The criteria are described below:
  Roeleveld et al. (1996): Score 11 - Restoration present, defect at the margin and/or wear of the surface; > 0.5 mm in depth, repair needed; Score 12 - Restoration present; underfilled > 0.5 mm, no gap, repair needed; Score 13 - Restoration overfilled > 0.5 mm, repair needed; Score 30 - Restoration not present, bulk fracture, loose, (partly) lost; repair needed (if still possible without exposing the pulp).
  Frencken et al. (2006): Score 2 - Restoration present, marginal defect between 0.5mm and 1.0 mm, repair needed. Score 3 - Restoration present, marginal defect between > 1.0 mm, repair needed.
Necessity to repair the restoration | 24 months.
  The necessity to repair the evaluated restorations during the follow-up examinations will be assessed by the Roeleveld et al. (1996) criteria (scores 11, 12, 13 and 30) or Frencken et al. (1996) criteria (scores 2 and 3). The criteria of the respective scores are described below:
  Roeleveld et al. (1996) Score 11 - Restoration present, defect at the margin and/or wear of the surface; > 0.5 mm in depth, repair needed. Score 12 - Restoration present; underfilled > 0.5 mm, no gap, repair needed. Score 13 - Restoration overfilled > 0.5 mm, repair needed. Score 30 - Restoration not present, bulk fracture, loose, (partly) lost; repair needed (if still possible without exposing the pulp). Frencken et al. (2006) Score 2 - Restoration present, marginal defect between 0.5mm and 1.0 mm, repair needed. Score 3 - Restoration present, marginal defect between > 1.0 mm, repair needed.
Restoration replacement | 24 months.
  Necessity of restoration replacement due to restoration loss (total or partial), with no signs of pulp involvement. For restorations involving occlusal surfaces, score 4 of Frencken et al. criteria (1996) will be considered. For restorations involving other surfaces, the scores 21, and 30.
Presence of secondary caries lesion with dentin exposure | 24 months.
  Caries lesion with dentin exposure around evaluated restorations detected in the follow-up examinations will be assessed by the Roeleveld et al. criteria (scores 20 and 21). The criteria of the respective scores are described below:
  Score 20 - Secondary caries, discoloration in depth, surface hard and intact, caries within dentin; repair needed. Score 21 - Secondary caries. Surface defect, caries within dentin; repair needed. Frencken criteria system does not deal with this aspect. Therefore, we considered the same parameters described above
Restored teeth that presents symptoms of pulp inflammation or episode of pain | 24 months.
  The restored teeth that presents symptoms of pulp inflammation or episode of pain during the follow-up examinations and need to be extracted will be assessed by the Roeleveld et al. criteria (score 40) for all types of restorations. The criteria of the respective score is described below:
  Score 40 - Inflammation of the pulp (restoration still in situ, not categorized in the former categories); fistula or severe pain complaints; extraction needed.

OTHER OUTCOMES:
Impact of Oral Health on quality of life | 24 months
  Impact of Oral Health on quality of life of the children participants in the study will be assessed through the questionnaire "Early Childhood Oral Health Impact Scale" (ECOHIS). The questionnaire is answered by the parents and contains 13 questions, divided into two sections: a child impact section with 4 domains (child symptoms, function, psychological, and self-image/social interaction domains) and a family impact section with 2 domains (parental distress and family function). Respondents answer the questions using a rating scale from 0 to 5, and total scores can range from 0 to 52. Score r corresponds to the "don't know" answer. Higher ECOHIS scores are indicative of greater negative impacts of oral health problems on quality of life. The questionnaire will be applied at the baseline and after 24 months of follow-up, preferentially to the same parent who responded the first questionnaire.
Cost of the treatments | 24 months
  The cost of the treatments performed during the follow-up per child considering the teeth included in our sample.

CONTACTS AND LOCATIONS:
Overall Officials: Fausto M Mendes, PhD, Principal Investigator — School of Dentistry, University of Sao Paulo
Locations (1):
- School of Dentistry, University of Sao Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Ismail AI, Pitts NB, Tellez M; Authors of International Caries Classification and Management System (ICCMS); Banerjee A, Deery C, Douglas G, Eggertsson H, Ekstrand K, Ellwood R, Gomez J, Jablonski-Momeni A, Kolker J, Longbottom C, Manton D, Martignon S, McGrady M, Rechmann P, Ricketts D, Sohn W, Thompson V, Twetman S, Weyant R, Wolff M, Zandona A. The International Caries Classification and Management System (ICCMS) An Example of a Caries Management Pathway. BMC Oral Health. 2015;15 Suppl 1(Suppl 1):S9. doi: 10.1186/1472-6831-15-S1-S9. Epub 2015 Sep 15. No abstract available. PMID 26391116
- [Background] Hickel R, Peschke A, Tyas M, Mjor I, Bayne S, Peters M, Hiller KA, Randall R, Vanherle G, Heintze SD. FDI World Dental Federation - clinical criteria for the evaluation of direct and indirect restorations. Update and clinical examples. J Adhes Dent. 2010 Aug;12(4):259-72. doi: 10.3290/j.jad.a19262. PMID 20847997
- [Background] Martins-Junior PA, Ramos-Jorge J, Paiva SM, Marques LS, Ramos-Jorge ML. Validations of the Brazilian version of the Early Childhood Oral Health Impact Scale (ECOHIS). Cad Saude Publica. 2012 Feb;28(2):367-74. doi: 10.1590/s0102-311x2012000200015. PMID 22331162
- [Background] Shivakumar K, Prasad S, Chandu G. International Caries Detection and Assessment System: A new paradigm in detection of dental caries. J Conserv Dent. 2009 Jan;12(1):10-6. doi: 10.4103/0972-0707.53335. PMID 20379434
- [Background] Roeleveld AC, van Amerongen WE, Mandari GJ. Influence of residual caries and cervical gaps on the survival rate of Class II glass ionomer restorations. Eur Arch Paediatr Dent. 2006 Jun;7(2):85-91. doi: 10.1007/BF03320820. PMID 17140533
- [Derived] Olegario IC, Moro BLP, Tedesco TK, Freitas RD, Passaro AL, Garbim JR, Oliveira R, Mendes FM; CARDEC 03 collaborative group; Raggio DP. Use of rubber dam versus cotton roll isolation on composite resin restorations' survival in primary molars: 2-year results from a non-inferiority clinical trial. BMC Oral Health. 2022 Oct 10;22(1):440. doi: 10.1186/s12903-022-02449-y. PMID 36217147
- [Derived] Moro BLP, Pontes LRA, Maia HC, Freitas RD, Tedesco TK, Raggio DP, Braga MM, Ekstrand KR, Imparato JCP, Cenci MS, Mendes FM. Clinical Accuracy of Two Different Criteria for the Detection of Caries Lesions around Restorations in Primary Teeth. Caries Res. 2022;56(2):98-108. doi: 10.1159/000523951. Epub 2022 May 3. PMID 35504257
- [Derived] Freitas RD, Moro BLP, Pontes LRA, Maia HCM, Passaro AL, Oliveira RC, Garbim JR, Vigano MEF, Tedesco TK, Deery C, Raggio DP, Cenci MS, Mendes FM, Braga MM; CARDEC collaborative group - CARDEC-03 trial. The economic impact of two diagnostic strategies in the management of restorations in primary teeth: a health economic analysis plan for a trial-based economic evaluation. Trials. 2021 Nov 12;22(1):794. doi: 10.1186/s13063-021-05722-7. PMID 34772437
- [Derived] Moro BLP, Signori C, Freitas RD, Pontes LRA, Lenzi TL, Tedesco TK, Raggio DP, Braga MM, Ekstrand KR, Cenci MS, Mendes FM; CARDEC collaborative group; CaCIA collaborative group. The effect of two clinical criteria in the assessment of caries lesions around restorations in children (CARDEC-03): study protocol for a diagnostic randomized clinical trial. F1000Res. 2020 Jun 26;9:650. doi: 10.12688/f1000research.23801.3. eCollection 2020. PMID 33520191